CLINICAL TRIAL: NCT05135169
Title: Multi-organ Transit Time Acquisition Using Contrast Ultrasound
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ken Monahan, Assistant Professor, Vanderbilt University Medical Center
Other Study IDs: IRB 212087
Record Dates: First submitted 2021-11-02; First posted 2021-11-26 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Contrast administration
  Interventions: Drug: Definity Suspension for Injection

INTERVENTIONS:
Drug: Definity Suspension for Injection — Administration of Definity

SUMMARY:
Echocardiographic contrast will be administered to volunteers for the purpose of measuring transit time through various organs/vascular beds

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* able to give informed consent

Exclusion Criteria:

1. Known allergic reaction to Definity ultrasound contrast
2. Pregnancy/Nursing - as assessed/disclosed by the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cross-section of VHVI faculty and sonographers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
transit time | during procedure
  time it takes for contrast to traverse an organ

CONTACTS AND LOCATIONS:
Locations (1):
- VUMC, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No